CLINICAL TRIAL: NCT02779075
Title: Exendin-9,39 and Satiety After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Principal Investigator, Adrian Vella, MD, FRCP (Edin), Consultant Division or Endocrinolgy, Diabetes and Nutrition, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16-001973
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Sleeve Gastrectomy; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): 0.9% NaCL (saline) intravenously for 6 hours.
  Interventions: Drug: Saline
- Exendin-9,39 (Active Comparator): Exendin-9,39 intravenously for 6 hours.
  Interventions: Drug: Exendin-9,39

INTERVENTIONS:
Drug: Saline — Subjects will be studied on 2 occasions, in random order. During the saline study they will be infused with saline.
  Arms: Saline
Drug: Exendin-9,39 — Subjects will be studied on 2 occasions, in random order. During the Exendin-9,39 study day they will be infused with Exendin-9,39. Exendin-9,39 blocks the actions of specific hormones called incretins, that are produced in the gut in health and in larger quantities after gastric bypass surgery.
  Arms: Exendin-9,39

SUMMARY:
The overall aim of the application is to determine the contribution of the elevated incretin hormone concentrations seen after certain types of bariatric surgery to the regulation of food intake and satiety.

DETAILED DESCRIPTION:
Both Sleeve Gastrectomy (SG) and Roux-en-Y Gastric Bypass (RYGB) increase GLP-1 concentrations, although this is of lesser magnitude in SG compared to RYGB. Data suggests that endogenous GLP-1 is at least partially responsible for reducing free-choice caloric intake after RYGB, providing a mechanism underlying differences between procedures. Inhibition of GLP-1 action with Exendin-9,39 after RYGB accelerates gastric emptying. These observations suggest that factors other than anatomy regulate the upper gastrointestinal response to food ingestion. It is therefore reasonable to consider that the postprandial rise in GLP-1 might affect feeding behavior after RYGB, and to a lesser extent SG, where the increase in GLP-1 is less marked.

ELIGIBILITY:
Inclusion Criteria:

* Undergone either sleeve gastrectomy or Roux-en-Y Gastric Bypass surgery within prior 2 years
* Healthy, with no active systemic illness

Exclusion Criteria:

* Pregnancy
* Functional or organic bowel symptoms
* Systemic illness
* Diabetes
* Bariatric surgery > 2 years

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kittah E, Camilleri M, Jensen MD, Vella A. A Pilot Study Examining the Effects of GLP-1 Receptor Blockade Using Exendin-(9,39) on Gastric Emptying and Caloric Intake in Subjects With and Without Bariatric Surgery. Metab Syndr Relat Disord. 2020 Nov;18(9):406-412. doi: 10.1089/met.2020.0049. Epub 2020 Aug 20. PMID 32833560

RESULTS

PARTICIPANT FLOW:
Groups:
- First Saline Then Exendin-9,39: First Intervention (Day 1 (6 hours of saline infusion) during which a test meal and a free-choice buffet meal were consumed, Washout (14 days), and the Second Intervention Day 16 (6 hours of Exendin-9,39 infusion) during which a test meal and a free-choice buffet meal were consumed.
- First Exendin-9,39 Then Saline: First Intervention (Day 1 (6 hours of Exendin-9,39 infusion) during which a test meal and a free-choice buffet meal were consumed, Washout (14 days), and the Second Intervention Day 16 (6 hours of saline infusion) during which a test meal and a free-choice buffet meal were consumed.
Period: Overall Study
Arm/Group | First Saline Then Exendin-9,39 | First Exendin-9,39 Then Saline
Started | 16 | 13
Completed | 14 | 10
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — IV lost during 2nd study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cross-over Design: Subjects will be studied on 2 occasions, in random order.
  During the Exendin-9,39 study day they will be infused with Exendin-9,39. Exendin-9,39 blocks the actions of specific hormones called incretins, that are produced in the gut in health and in larger quantities after gastric bypass surgery.
  During the Saline study day they will be infused with saline as a control
Arm/Group | Cross-over Design
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Caloric Intake
Description: caloric intake from a free choice buffet within 5 hours after ingestion of a standard meal
Time Frame: 5 hours
Population: Analysis was confined to participants who did not withdraw consent after screening
Measure: Mean (Standard Error); unit: calories
Arm/Group | First Saline Then Exendin-9,39 | First Exendin-9,39 Then Saline
Number analyzed (Participants) | 16 | 13
calories
  Saline infusion | 531 (71) | 465 (107)
  Exendin-9,39 infusion | 444 (65) | 494 (98)

2. Secondary Outcome: Gastrointestinal Transit Measured Using Scintigraphy
Description: Time taken to empty 50% of stomach contents (GE50) measured using scintigraphy over the 4 hours after ingestion of a labeled meal
Time Frame: 4 hours
Population: Analysis was confined to participants who did not withdraw consent after screening
Measure: Mean (Standard Error); unit: minutes
Arm/Group | First Saline Then Exendin-9,39 | First Exendin-9,39 Then Saline
Number analyzed (Participants) | 16 | 13
minutes
  Saline infusion | 63 (13) | 48 (14)
  Exendin-9,39 infusion | 100 (24) | 141 (43)

ADVERSE EVENTS:
Time Frame: duration of experiment i.e 6 hours
Arm/Group | Saline | Exendin-9,39
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline (N=24) | Exendin-9,39 (N=24)
infiltration of intravenous line (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT02779075/Prot_SAP_000.pdf